CLINICAL TRIAL: NCT00001078
Title: An Observational Study of the Rate of Opportunistic Infection Events in HIV-Infected Children Who Have Demonstrated Immunologic Reconstitution and Who Have Discontinued OI Prophylaxis
Brief Title: A Study on the Rate of Opportunistic (AIDS-Related) Infections Among HIV-Positive Children Who Have Stopped Taking Their OI Preventive Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Purpose: Treatment
Other Study IDs: ACTG P1008; PACTG P1008
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: Viral Vaccines; AIDS-Related Opportunistic Infections; Anti-HIV Agents; Hepatitis A Virus, Human
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Hepatitis | interventions — Hepatitis A Vaccines

INTERVENTIONS:
Biological: Hepatitis A Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to find out if it is safe for HIV-positive children who are responding well to their anti-HIV treatment to stop taking medications that prevent AIDS-related infections (opportunistic infections) such as pneumonia and other bacterial infections. This is an observational study, meaning children will only be monitored to see if they develop any infections.

Children have been receiving medications to prevent complications of HIV infection, such as Pneumocystis carinii pneumonia (PCP), Mycobacterium avium complex (MAC) disease, or other bacterial infections. It is common for HIV-positive patients with low CD4 counts to receive these preventive medications. However, these drugs can have serious side effects, they are expensive, and it is possible for bacteria resistant to the drugs to grow. For these reasons, it may be beneficial to the child to stop taking these preventive medications if he/she has been on anti-HIV (antiretroviral) therapy and has improved CD4 counts. This study will look at how many children who stop taking their medications develop opportunistic infections.

DETAILED DESCRIPTION:
Due to the strong correlation between a significant decrease in CD4 count and the frequency and magnitude of OIs such as Pneumocystis carinii pneumonia (PCP), Mycobacterium avium complex (MAC), and severe bacterial infections, CD4 count has become the major criterion for initiating antimicrobial prophylaxis for OIs. However, despite the benefits of these antimicrobial drugs, all are associated with adverse side effects, and patients with reconstituted immune systems following antiretroviral therapy may be receiving prophylaxis unnecessarily. Benefits to stopping prophylaxis include: (1) elimination of adverse effects from drugs; (2) reduction in drug costs; and (3) removal of selective pressure for the development of drug-resistant microbes. These benefits must be weighed against the disadvantages, however, such as more frequent determinations of CD4 counts to assure maintenance of immunocompetence, more frequent occurrence of serious OIs otherwise preventable with prophylaxis in patients lost to follow-up, and possible occurrence of atypical PCP because of prior exposure to anti-PCP drugs. [AS PER AMENDMENT 04/26/02: The extent of complete immune restitution has not yet been defined. An important corollary of an incomplete immune recovery is that vaccination schedules might need to be adjusted to obtain optimal responses in HIV-infected patients on highly active antiretroviral therapy (HAART). Therefore, a third dose of hepatitis A virus vaccine will be administered.]

After pre-entry and entry laboratory studies, patients are followed every 8 weeks until the last patient has completed 104 weeks of study observation. Hepatitis A vaccination is administered at entry and Week 24 to measure responses to neoantigen. [AS PER AMENDMENT 04/26/02: All patients (except those co-enrolled in P1024 on or after November 1, 2001) who have received 2 doses of hepatitis A virus vaccine during the study will be offered an opportunity to enroll in Step II of P1008. Patients in Step II receive a third dose of hepatitis A vaccination at Week 104 or later. Additional blood samples are taken 8 weeks later for antibody detection and peripheral blood mononuclear cell (PBMC) cryopreservation.] All serious bacterial infections that are Grade 3 or higher and OI events are recorded and compared to historical event rates. Virologic and immunologic marker studies are done in all patients and correlated with the risk of developing serious bacterial infections or OI events. Patients are considered to have reached an endpoint if they develop PCP, 2 serious bacterial infections, other Category C OI diagnoses, or CD4% less than 15% and re-initiation of PCP prophylaxis.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 percent greater than or equal to 25 percent if they are under 6 years of age, or have a CD4 percent greater than or equal to 20 percent on 2 occasions if they are between the ages of 6 and 21.
* Have been receiving preventive treatment for PCP for at least 6 months and have not stopped treatment for more than 3 months before study entry.
* Are willing to stop taking preventive treatment for PCP and MAC.
* Have received the same continuous antiretroviral (anti-HIV) therapy for the 16 weeks before beginning the study. (Continuous therapy means missing no more than a total of 3 weeks during the 16 weeks.)
* Are between the ages of 2 and 21 years (consent of parent or guardian is required if under 18).

Exclusion Criteria

Children will not be eligible for this study if they:

* Have PCP.
* Have any other active infection, such as tuberculosis or toxoplasmosis, or any other significant disease.
* Are receiving chemotherapy for cancer or certain other medications.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Primary Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Dankner, Study Chair; Ram Yogev, Study Chair; Walter Hughes, Study Chair
Locations (50):
- United States (47):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Yale Univ Med School, New Haven, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Result] Weinberg A, Huang S, Fenton T, Patterson-Bartlett J, Gona P, Read JS, Dankner WM, Nachman S; IMPAACT P1008 Team. Virologic and immunologic correlates with the magnitude of antibody responses to the hepatitis A vaccine in HIV-infected children on highly active antiretroviral treatment. J Acquir Immune Defic Syndr. 2009 Sep 1;52(1):17-24. doi: 10.1097/QAI.0b013e3181b011f6. PMID 19617848